CLINICAL TRIAL: NCT04751942
Title: Post-operative Comparison Between Standard Gradient Compression Dressing vs. Non-Compressive Bioactive Garment on Pain, Swelling and Range of Motion Following Total Knee Arthroplasty
Brief Title: Reparel Knee Sleeve vs. TED Hose for Post-op Swelling, Pain and Range of Motion After Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Rachael Kilkenny, Orthopedic Program Coordinator, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20210037
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Results first posted 2025-11-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Osteoarthritis Knees Both
Keywords: post-operative swelling; total knee arthroplasty; TKA; TED hose; photobiomodulation
MeSH Terms: interventions — Stockings, Compression

STUDY DESIGN:
Intervention Model Description: prospective randomized control cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Non-compressive Bioactive Garment (Experimental): The non-compressive bioactive garment is a commercially available garment that is designed to reflect infrared waves generated by the wearer back into the soft tissue surrounded by the garment. The reflection of the infrared waves is intended to improve pain and swelling at the site. Patients following Total knee replacement are intended to wear morning and night for the first 2 weeks post-operatively, and then as tolerated for 4 weeks afterwards. The patients will then discontinue use of the sleeve after 6 weeks.
  Interventions: Device: Non-compressive Bioactive Garment
- Thrombo-Embolic Deterrent (Active Comparator): a gradient compression stocking that is currently the gold standard for deterring thromboembolic events and assisting with post-operative swelling after total knee replacements. Patients following Total knee replacement are intended to wear the TED hose morning and night for the first 2 weeks post-operatively, and then as tolerated for 4 weeks afterwards. The patients will then discontinue use of the sleeve after 6 weeks.
  Interventions: Device: thrombo-embolic deterrent

INTERVENTIONS:
Device: Non-compressive Bioactive Garment — patients will be assigned to wear the non-compressive bioactive garment following total knee arthroplasty
  Arms: Non-compressive Bioactive Garment
Device: thrombo-embolic deterrent — patients will be randomized to wear the gold standard TED hose following total knee arthroplasty
  Other Names: TED hose
  Arms: Thrombo-Embolic Deterrent

SUMMARY:
This prospective study will evaluate pain, swelling, ROM as well as narcotic use in post-operative total knee arthroplasty patients using novel Non-Compressive Bioactive Garment (NCBG) versus current standard of care gradient compression stocking (Thrombo-Embolic-Deterrent or TED hose). If NCBG proves to be more effective in these outcome areas, it will provide a new and comfortable way to reduce patient pain and swelling immediately following surgery

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is one of the most popular surgical procedures today. It is designed and proven to effectively reduce pain caused by end-stage osteoarthritis. Despite its achievements, up to 25% of patients remain dissatisfied after the procedure due to lingering pain, amongst other complaints. Post-operative swelling of the knee and leg is thought to be a contributor to this persistent pain.

Traditionally, a standard gradient compression stocking is applied to the knee and leg after surgery to reduce this pain and swelling. However, due to ineffectiveness or patient non-compliance, compression stockings are often not entirely successful at preventing edema. The recently developed NCPS is a lower extremity garment comprised of a technical fabric that is thought to be able to prevent edema and reduce pain all in a comfortable, user-friendly manner. The purpose of this study is to determine if the NCPS is effective at improving post-operative pain, swelling, ROM and analgesic use associated with TKA.

Pain and prolonged recovery time associated with post-operative swelling are two factors that contribute to patient dissatisfaction following TKA. Swelling of the knee following TKA is caused by intraarticular bleeding and inflammation of the periarticular tissues, which can lead to a decrease in functional performance including pain and delayed rehabilitation. In a study by Noble et al, 1/3 of dissatisfied patients reported that their knees swelled at least once per week, leading to pain and discomfort1. Decreased quadriceps strength following knee surgery has been shown to prolong recovery1-8. Fahrer et al showed that knee effusions inhibited reflex neurons and altered kinetics and muscle activity in quadriceps, which ultimately causes decreased strength2. Holm et al later showed us that knee swelling played a part in post-operative quadriceps strength following TKA3. Ultimately, if post-operative swelling can effectively be reduced, patient recovery could be expedited and patient satisfaction could be improved.

Compression stockings have been utilized to attempt to reduce post-operative swelling. Compression works to prevent swelling by reducing the hydrostatic pressure in the leg. Reducing hydrostatic pressure prevents the capillaries from oozing and allows blood to move freely from the superficial to the deep venous system, subsequently allowing excess fluid to flow away from the interstitial space9.

More recently, the use of gradient compression stocking following TKA has come into question for its efficacy. While the application of external pressure from these gradient compression stocking is beneficial for a period, they are often unable to exert a sufficient amount of pressure long enough to prevent painful edema for an extended amount of time. A study by Bowling et al showed that these garments showed sufficient compression during the first few hours after surgery, but the pressure they applied dropped with time and required daily measurements and refitting to maintain appropriate and therapeutic compression10. This poses a problem not only medically, but financially as well. These compression stockings lose their fit so quickly, new ones must be prescribed frequently, leading to costly bills for the patient. It's clear that compression stockings are not as effective as once thought when it comes to controlling pain and swelling post-operatively.

A potential solution to the problems posed by traditional compression stocking is the NCPG. The garment is comprised of a semi-conductive material ground to nanoparticles that are embedded into the fibers, formed into a three-dimensional woven fabric for optimized comfort. Instead of relying on compression, NCPS utilizes the body's own thermal energy to generate infrared energy. The infrared energy generated is reflected back at the body and modifies cellular activity at the level of the mitochondria through a process known as photobiomodulation14-15. This process of photobiomodulation is hypothesized to improve swelling and tissue healing by increasing the activity of mitochondria and the availability of cellular energy in the form of ATP.

This study seeks to determine if NCPS use of infrared energy is more successful at reducing pain and swelling following TKA than traditional gradient compression dressing.

We will enroll 100 subjects throughout all sites involved in the study.

Patients will be recruited in the office setting after all non-operative modalities for controlling pain associated with end-stage osteoarthritis of the knee have been exhausted. Patients will then be presented with the option of total knee replacement. After patient has agreed to undergo TKA, patients will then be asked (in a face-to-face setting) if they would like to participate in the study.

Patients will be approached in the office setting after it has been determined that they have failed conservative management of advanced knee arthritis. Patients will be in the surgeons' clinic behind closed doors with the performing surgeon and potentially other members of the research team. Consent will be obtained in the office after scheduling total knee arthroplasty procedure. The consent process is expected to take 30 minutes, but more time is available to ensure that patients have all their questions answered prior to signing the consent form.

Patients will be enrolled in study prior to surgery, outlined above in the consent process.

On the day of surgery, patients will arrive and will be situated in the pre-operative holding area. A trained member of the research team will meet the patient in the pre-operative holding area and will measure the circumference of the patient's leg at the mid-thigh, mid-knee and mid-calf. The patient's range of motion of the operative leg will be measured in flexion and extension. All measurements will be recorded in redcap.

The patient will then go on to have their primary total knee arthroplasty by standard of care procedure. Both cruciate retaining and posterior stabilized total knee replacement designs will be included in the study. Following closure of the surgical site and placement of a post-operative occlusive dressing, the operative leg will be measured once more for circumference and range of motion, and the values will be entered into redcap. The patient will then be placed in their randomized post-operative sleeve/device and will be transferred to the PACU and will receive the standard post-operative treatment.

On post-operative day one, patient's will be seen and evaluated in their inpatient rooms. Their leg measurements will be taken again with the knee sleeve/compressive gradient dressing pulled down. Patient's skin will be inspected for any reactions to the sleeve and a standard post-operative examination will be performed to ensure no neurovascular compromise, blood clots, infections or other post-operative complications.

Patients will likely be discharged on post-operative day 1. Patients that have not been discharged on post-operative day 1 will not be measured on post-operative day 2.

Patients will be provided with a journal that they will use every daily to track their pain based on a visual analog scale and their narcotic consumption (number of Percocet or tramadol pills). Patients will also use their journal to log the number of hours they wore their sleeve each day. Patients will continue to log the number of pain medications taken and hours wearing the sleeve for 6 weeks

Sleeves will be worn morning and night removing them only for hygiene and washing of sleeve for 2 weeks. After 2 weeks, the patient's will wear the sleeve as much as they can tolerate day and night. At 6 weeks, sleeves will be discontinued all together. Final ROM and Circumference Measurements will be obtained at 12 weeks post-operative mark.

Patients will be asked to fill out the Knee Society Score questionnaire at the time of consent and at each post-operative visit.

The Reparel leg sleeve is the experimental device being investigated in this study. It is intended to improve swelling in the post-operative knee.

Allscripts Electronic Medical Records will be used to collect data about patients during their inpatient, post-operative stay. UH Care ambulatory EMR and Medent EMR will be used in the outpatient setting to collect data and track post-operative clinic visits.

The enrollment period will be 1 year from the time of the first patient enrolled in the study. The enrollment period may be expanded to allow for the investigators to reach their goal of 100 patients. The total amount of time each patient will be involved in the study will be 12 weeks. Patients will only be required to wear the post-operative sleeve/dressing for 6 weeks post-operatively. Patients will continue to record their narcotic consumption and pain scores for 12 weeks post-operatively

Date to be collected:

Mid-thigh, mid-knee, and mid-calf measurements ROM measurements in knee flexion and knee extension Visual analog Pain scale Knee society score (KSS) Narcotic consumption Name Medical record number Surgeon weight

Data Analysis Plan:

Demographics will be reported using descriptives such as count data and percentages. Differences between groups at baseline (pre-op) will be reported using two-tailed independent t-tests for continuous variables, and chi-square or Fisher's Exact tests for categorical data, as appropriate.

The primary outcomes of range of motion, leg circumference, and pain ratings will be compared post-op between conditions using two-tailed independent t-tests. Should clinically relevant demographics differ significantly between conditions pre-op (baseline), post-op comparisons will instead be conducted using one-way ANCOVAs controlling for differences at pre-op (baseline). These comparisons will additionally be made at multiple additional time-points throughout a 12-week post-op time period.

A priori power analyses were calculated for two-tailed independent t-tests for each primary outcome, using an alpha of .05, power = .80. Each of these are reported and the average of these numbers is used to calculate the final sample size. Clinically significant reductions in pain are defined as a 2-point change with a standard deviation of 2.5 using a 10-point scale; 84 patients were estimated. Clinically significant changes in range of motion are defined as: 10 degrees of difference from a 0-140 degree estimated range of values. Clinically significant changes in leg circumference are defined as: 1 cm difference in leg circumference using a 15-30 estimated range of values. To identify medium effect sizes of .55, 106 patients were estimated. Averaging these values, 99 patients were estimated. To ensure equal numbers of patients in each condition, 100 patients will be recruited for this study.

The data will be monitored every 10 patients to assess for completeness, accuracy and adherence to the protocol. We will also be monitoring for any obvious safety concerns that may arise.

There will not be a designated safety team assigned.

ELIGIBILITY:
Inclusion Criteria:

* Primary unilateral Total Knee Replacement - Cruciate retaining and Posterior stabilized designs

Exclusion Criteria:

* Leg circumference > 23 in.
* Allergy to silicone/polyester
* Current DVT
* Primary Inflammatory Type arthritis (i.e. rheumatoid arthritis)
* Inability to follow standardized post op and rehab protocols
* Lymphedema
* History of Vascular Bypass Surgery on Operative Limb (i.e. Fem-Pop or Fem-Fem)
* Chronic Narcotic Use History

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachael A Kilkenney, MBA,BSN, Principal Investigator — University Hospitals
Locations (1):
- University Hospitals Beachwood Medical Center, Beachwood, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noble PC, Conditt MA, Cook KF, Mathis KB. The John Insall Award: Patient expectations affect satisfaction with total knee arthroplasty. Clin Orthop Relat Res. 2006 Nov;452:35-43. doi: 10.1097/01.blo.0000238825.63648.1e. PMID 16967035
- [Background] Fahrer H, Rentsch HU, Gerber NJ, Beyeler C, Hess CW, Grunig B. Knee effusion and reflex inhibition of the quadriceps. A bar to effective retraining. J Bone Joint Surg Br. 1988 Aug;70(4):635-8. doi: 10.1302/0301-620X.70B4.3403614.
- [Background] Holm B, Kristensen MT, Bencke J, Husted H, Kehlet H, Bandholm T. Loss of knee-extension strength is related to knee swelling after total knee arthroplasty. Arch Phys Med Rehabil. 2010 Nov;91(11):1770-6. doi: 10.1016/j.apmr.2010.07.229. PMID 21044725
- [Background] Spencer JD, Hayes KC, Alexander IJ. Knee joint effusion and quadriceps reflex inhibition in man. Arch Phys Med Rehabil. 1984 Apr;65(4):171-7. PMID 6712434
- [Background] Hopkins JT, Ingersoll CD, Krause BA, Edwards JE, Cordova ML. Effect of knee joint effusion on quadriceps and soleus motoneuron pool excitability. Med Sci Sports Exerc. 2001 Jan;33(1):123-6. doi: 10.1097/00005768-200101000-00019. PMID 11194097
- [Background] McNair PJ, Marshall RN, Maguire K. Swelling of the knee joint: effects of exercise on quadriceps muscle strength. Arch Phys Med Rehabil. 1996 Sep;77(9):896-9. doi: 10.1016/s0003-9993(96)90277-4. PMID 8822681
- [Background] Mizner RL, Petterson SC, Stevens JE, Vandenborne K, Snyder-Mackler L. Early quadriceps strength loss after total knee arthroplasty. The contributions of muscle atrophy and failure of voluntary muscle activation. J Bone Joint Surg Am. 2005 May;87(5):1047-53. doi: 10.2106/JBJS.D.01992. PMID 15866968
- [Background] Bowling K, Ratcliffe C, Townsend J, Kirkpatrick U. Clinical thromboembolic detterrent stockings application: are thromboembolic detterrent stockings in practice matching manufacturers application guidelines. Phlebology. 2015 Apr;30(3):200-3. doi: 10.1177/0268355514542843. Epub 2014 Jul 2. PMID 24990877
- [Background] Munk S, Jensen NJ, Andersen I, Kehlet H, Hansen TB. Effect of compression therapy on knee swelling and pain after total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2013 Feb;21(2):388-92. doi: 10.1007/s00167-012-1963-0. Epub 2012 Mar 28. PMID 22453307
- [Background] Ross M, Worrell TW. Thigh and calf girth following knee injury and surgery. J Orthop Sports Phys Ther. 1998 Jan;27(1):9-15. doi: 10.2519/jospt.1998.27.1.9. PMID 9440035
- [Background] Smith J, Stevens J, Taylor M, Tibbey J. A randomized, controlled trial comparing compression bandaging and cold therapy in postoperative total knee replacement surgery. Orthop Nurs. 2002 Mar-Apr;21(2):61-6. doi: 10.1097/00006416-200203000-00009. PMID 11949239
- [Background] de Freitas LF, Hamblin MR. Proposed Mechanisms of Photobiomodulation or Low-Level Light Therapy. IEEE J Sel Top Quantum Electron. 2016 May-Jun;22(3):7000417. doi: 10.1109/JSTQE.2016.2561201. PMID 28070154
- [Background] Karu TI. Mitochondrial signaling in mammalian cells activated by red and near-IR radiation. Photochem Photobiol. 2008 Sep-Oct;84(5):1091-9. doi: 10.1111/j.1751-1097.2008.00394.x. Epub 2008 Jul 18. PMID 18651871

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-compressive Bioactive Garment | Thrombo-Embolic Deterrent
Started | 14 | 9
Completed | 5 | 3
Not Completed | 9 | 6
Not completed — Lost to Follow-up | 9 | 6

BASELINE CHARACTERISTICS:
Population: Baseline data collection was impacted by workflow transitions and adjustments during the study, making reporting baseline data impossible. During the study period, transcription errors lead to missing data elements. Measures were taken since implementation to reinforce consistency in the data capture practices to ensure outcome measure data was consistent, however baseline data was left out and therefore not able to be reported.
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-compressive Bioactive Garment | Thrombo-Embolic Deterrent | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Change in Leg Circumference (cm)
Description: circumference of the leg will be measured pre-operatively, immediately post operatively, and at regular intervals post-operatively.
Time Frame: Preop, 2 weeks post op, 6 weeks post-op, 3 months post-op
Population: Data was collected for participants that showed at each follow up apt, some did not come to all follow up apts.
Measure: Mean (Standard Deviation); unit: Leg circumference (cm)
Arm/Group | Non-compressive Bioactive Garment | Thrombo-Embolic Deterrent
Number analyzed (Participants) | 13 | 8
Leg circumference (cm)
  Pre-op | 44.06 (3.77) | 44.77 (6.34)
  2 weeks Post-op: number analyzed (Participants) | 12 | 8
  2 weeks Post-op | 44.18 (4.25) | 49.99 (5.19)
  6 weeks Post-op: number analyzed (Participants) | 8 | 3
  6 weeks Post-op | 45.17 (5.85) | 46.14 (2.16)
  3 months Post-op: number analyzed (Participants) | 5 | 3
  3 months Post-op | 46.36 (5.65) | 45.89 (1.87)

2. Primary Outcome: Change in Pain Score (1-10)
Description: patient's subjective pain scores will be recorded daily in a pain journal using a visual analog scale from 1-10, values are grouped into mild (1-3), moderate (4-6), and severe (7-10) pain.
Time Frame: Pre-op, 1 week Post-op, 2 weeks Post-op, 6 weeks Post-op, 3 months Post-op
Population: Data was collected for participants that showed at each follow up apt, some did not come to all follow up apts.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-compressive Bioactive Garment | Thrombo-Embolic Deterrent
Number analyzed (Participants) | 14 | 9
score on a scale
  Pre-op | 4.07 (1.8) | 4.44 (1.64)
  1 week Post-op: number analyzed (Participants) | 9 | 5
  1 week Post-op | 3.67 (1.25) | 4 (1.67)
  2 weeks Post-op: number analyzed (Participants) | 12 | 8
  2 weeks Post-op | 2.92 (1.5) | 4.25 (2.44)
  6 weeks Post-op: number analyzed (Participants) | 8 | 3
  6 weeks Post-op | 1.25 (0.97) | 2 (0.82)
  3 months Post-op: number analyzed (Participants) | 5 | 3
  3 months Post-op | 1.4 (0.8) | 1.33 (0.47)

3. Primary Outcome: Change in Range of Motion
Description: patients passive flexion range of motion will be tested pre-operatively, immediately post-operatively, and at regular intervals post-operatively
Time Frame: Pre-op, 2 weeks Post-op, 6 weeks Post-op, 3 months Post-op
Population: Data was collected for participants that showed at each follow up apt, some did not come to all follow up apts.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Non-compressive Bioactive Garment | Thrombo-Embolic Deterrent
Number analyzed (Participants) | 13 | 8
Degrees
  Pre-op | 121.85 (13.81) | 116.88 (25.61)
  2 weeks Post-op: number analyzed (Participants) | 12 | 7
  2 weeks Post-op | 99.08 (13.16) | 95.29 (15.46)
  6 weeks Post-op: number analyzed (Participants) | 8 | 3
  6 weeks Post-op | 117.13 (15.91) | 114 (13.59)
  3 months Post-op: number analyzed (Participants) | 5 | 3
  3 months Post-op | 113.4 (5.12) | 115.33 (7.76)

4. Primary Outcome: Change in Narcotic Consumption
Description: the narcotic consumption in Milligrams of morphine equivalents (MME) per day will be recorded post-operatively while in the hospital and will be self reported by the patient in a journal as "number of pills" taken
Time Frame: 1 week Post-op, 2 weeks Post-op. 6 weeks Post-op, 3 months Post-op
Population: Data was collected for participants that showed at each follow up apt, some did not come to all follow up apts.
Measure: Mean (Standard Deviation); unit: Milligrams of morphine equivalents.day
Arm/Group | Non-compressive Bioactive Garment | Thrombo-Embolic Deterrent
Number analyzed (Participants) | 12 | 8
Milligrams of morphine equivalents.day
  1 week Post-op: number analyzed (Participants) | 9 | 5
  1 week Post-op | 1.56 (1.42) | 2 (1.79)
  2 week Post-op | 1.58 (1.26) | 2.5 (2.35)
  6 weeks Post-op: number analyzed (Participants) | 8 | 3
  6 weeks Post-op | 0.25 (0.43) | 0 (0)
  3 months Post-op: number analyzed (Participants) | 5 | 8
  3 months Post-op | 0 (0) | 0 (0)

5. Primary Outcome: Change in Knee Society Score (KSS)
Description: a validated system that combines an objective physician-derived component with a subjective patient-derived component that evaluates pain relief, functional abilities, satisfaction, and fulfillment of expectations. Patients will fill out this questionnaire pre-operatively and at each post-operative visit. With lower scores indicating lower pain/difficulty with daily activities and higher scores indicating higher pain/difficulty with daily activities.
Time Frame: Pre-op, 1 week Post-op, 2 weeks Post-op, 6 weeks Post-op, 3 months Post-op
Population: Data was collected for participants that showed at each follow up apt, some did not come to all follow up apts.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Non-compressive Bioactive Garment | Thrombo-Embolic Deterrent
Number analyzed (Participants) | 14 | 9
units on a scale
  Pre-op | 38.29 (16.25) | 40.33 (13.81)
  1 week Post-op: number analyzed (Participants) | 9 | 5
  1 week Post-op | 33.33 (14.45) | 33 (16.90)
  2 weeks Post-op: number analyzed (Participants) | 12 | 8
  2 weeks Post-op | 23.92 (14.30) | 31.25 (23.68)
  6 weeks Post-op: number analyzed (Participants) | 8 | 3
  6 weeks Post-op | 10.63 (8.01) | 15.67 (4.78)
  3 months Post-op: number analyzed (Participants) | 5 | 3
  3 months Post-op | 11.2 (7.96) | 22.67 (23.57)

ADVERSE EVENTS:
Time Frame: Up to 3 months post-op
Arm/Group | Non-compressive Bioactive Garment | Thrombo-Embolic Deterrent
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/14 | 2/9
Other Adverse Events (participants affected / at risk) | 0/14 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-compressive Bioactive Garment (N=14) | Thrombo-Embolic Deterrent (N=9)
Surgical site infection (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Limitations to this study included the mid-study employment change of Corey Barnett, who had served as a primary data collection specialist. In addition, a transition to a new electronic medical record system within the practice introduced added complexity in monitoring patients both pre- and postoperatively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT04751942/Prot_SAP_000.pdf